CLINICAL TRIAL: NCT01565187
Title: Development of a Psychosocial Assessment Database for Reconstructive Hand Transplantation
Status: Terminated | Type: Observational
Why Stopped: Due to lack of enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sheila G. Jowsey, MD, Assistant Professor of Psychiatry and Director of Transplant Psychiatry, Mayo Clinic
Other Study IDs: 12-001131
Record Dates: First submitted 2012-03-14; First posted 2012-03-28 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Arm Injuries
Keywords: Hand Transplantation
MeSH Terms: conditions — Arm Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens to be gathered and used for this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- hand transplant candidates: Participants enrolled will be asked to complete behavioral questionnaires.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Transplant Effects Questionnaire, Response Evaluation Measure, Patient Health Questionnaire, Generalized Anxiety Scale, Alcohol Use Disorders Test, Body Image Questionnaire, Quality of Life Uniscale, Scales of Psychosocial Well-Being, Sense of Coherence Scale.
  Other Names: Psychometric instruments

SUMMARY:
A prospective multicenter study utilizing standardized instruments for the psychological assessment of hand transplant candidates pre and post-transplant as well as those candidates excluded for transplantation.

DETAILED DESCRIPTION:
The semi-structured psychological interview describes the assessment of significant psychosocial characteristics and it is based on the psychosocial domains of the "Transplant Evaluation Rating Scale (TERS)" by Twillman and colleagues for evaluating organ transplant candidates. The interview guide was developed as a tool to guide clinicians through the interview process for hand transplant candidates. The protocol highlights issues that are specific for reconstructive hand transplantation and give clinicians an immediate understanding of what type of information is necessary to conduct a comprehensive psychosocial assessment.

Additionally, the psychological assessment provides standardized psychological screening procedures and continuous follow-up ratings by psychometrical testing. The test battery will be performed at the time of initial psychosocial assessment, immediately after transplant, at six and twelve months for the transplant candidates and at initial evaluation, six and twelve months for candidates excluded for transplant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Undergoing evaluation for hand transplantation

Exclusion Criteria:

* unable to complete surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Candidate who will be receiving a hand transplant at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-02; Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Assessment of change in Psychosocial characteristics of hand transplantation candidates | one year posttransplant
  Using validated psychometric instruments and description of psychosocial characteristics based on a standardized assessment instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Jowsey, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials